CLINICAL TRIAL: NCT02016950
Title: East Sussex Long-term Pacemaker Arrhythmia Analysis
Brief Title: Long-term Pacemaker Arrhythmia Analysis
Status: Completed | Type: Observational
Sponsor: Eastbourne General Hospital (Other)
Responsible Party: Principal Investigator, Neil Sulke, Consultant Cardiologist, Eastbourne General Hospital
Other Study IDs: ESHT Pacemaker analysis
Record Dates: First submitted 2013-12-11; First posted 2013-12-20 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Permanent pacemaker: Pre-existing permanent pacemakers

SUMMARY:
Investigators seek to observe the long term patterns of arrhythmias detected by permanent pacemakers.

ELIGIBILITY:
Inclusion Criteria:

* Pre-existing dual chamber permanent pacemaker

Exclusion Criteria:

* Nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those with permanent pacemakers
Sampling Method: Non-Probability Sample
Enrollment: 2551 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation burden | 28 days to 1 year
  Proportion of monitored time in atrial fibrillation

SECONDARY OUTCOMES:
Atrial fibrillation episode frequency | 28 days to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sulke, MD, Principal Investigator — Eastbourne General Hospital
Locations (1):
- Eastbourne General Hospital, Eastbourne, E Sussex, United Kingdom

REFERENCES:
- [Derived] Sugihara C, Veasey R, Freemantle N, Podd S, Furniss S, Sulke N. The development of AF over time in patients with permanent pacemakers: objective assessment with pacemaker diagnostics demonstrates distinct patterns of AF. Europace. 2015 Jun;17(6):864-70. doi: 10.1093/europace/euv032. PMID 26023175